CLINICAL TRIAL: NCT06947616
Title: Effect of Mild Therapeutic Hypothermia on the Doses of Vasopressors and Inotropes in Cardiogenic Shock Complicating Acute Myocardial Infarction: A Randomized Controlled Trial
Brief Title: Effect of Mild Therapeutic Hypothermia on the Doses of Vasopressors and Inotropes in Cardiogenic Shock Complicating Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrazek Abdelmonem Abdelaal, Resident of Cardiology Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33716/3/20
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Mild Therapeutic Hypothermia; Cardiogenic Shock; Acute Myocardial Infarction; Vasopressors; Inotropes
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild therapeutic hypothermia group (Experimental): Patients received mild therapeutic hypothermia (MTH) to 33°C for 24-36 h
  Interventions: Drug: Mild therapeutic hypothermia
- Control group (No Intervention): Patients did not receive mild therapeutic hypothermia (MTH)

INTERVENTIONS:
Drug: Mild therapeutic hypothermia — Patients received mild therapeutic hypothermia (MTH) to 33°C for 24-36 h
  Arms: Mild therapeutic hypothermia group

SUMMARY:
The study aimed to assess the effects of mild therapeutic hypothermia (MTH) on vasopressors and inotropes in patients with cardiogenic shock (CS) due to acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a condition characterized by a severe lack of blood flow to vital organs caused by primary malfunction of the heart, as described by the European Society of Cardiology (ESC) and the American Heart Association (AHA). Acute myocardial infarction (AMI) is a prevalent etiology of CS, constituting a minimum of 30% of the instances. 50% of CS cases manifest upon hospital admission, whereas the remaining 50% occur after hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Age from 50 to 70 years.
* Both sexes.
* Cardiogenic shock post AMI defined by systolic blood pressure <90 mm Hg for >30 minutes or motropes required to maintain a systolic blood pressure >90 mm Hg in the absence of hypovolemia with signs of pulmonary congestion and signs of impaired organ perfusion defined by at least 1 of the following: altered mental status; cold, clammy skin; urine output <30 mL/h; or arterial lactate >2 mmol/L.

  2. Intubated and sedated

Exclusion Criteria:

1. Self-ventilated
2. Indication for targeted temperature management by current guidelines "out of hospital cardiac arrest with return of spontaneous circulation (ROSC)"

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke | 30 day after the procedure
  Incidence of stroke until day 30 was recorded.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Up to 7 days
  Duration of mechanical ventilation was recorded.
Length of intensive care unit stay | Up to 2 weeks after the procedure
  Length of intensive care unit (ICU) stay refers to the total duration a patient remains in the ICU, beginning from the moment of admission to the ICU until their discharge or transfer to a less intensive care setting, such as a regular hospital ward or home.
Duration of inotropic support | Intraoperatively
  Duration of inotropic support was recorded.
Incidence of mortality | 30 days after the procedure
  Incidence of mortality was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author